CLINICAL TRIAL: NCT04708678
Title: Long-term Efficacy of Doppler Ligation With Mucopexy in the Treatment of Internal Hemorrhoidal Disease
Acronym: HEM_THD
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: HEM_THD
Record Dates: First submitted 2021-01-12; First posted 2021-01-14 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Hemorrhoids
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A classic distinction is made between internal and external hemorrhoidal pathology. External hemorrhoids can present with thrombosis, which causes painful swelling; internal hemorrhoids by rectal bleeding, prolapse, and more rarely thrombosis. Hemorrhoidal pathology is one of the most frequent reasons for consultation in proctology. Its prevalence is probably underestimated due to taboos and the frequent self-medication of patients, but it is considered high in the general population.

The therapeutic management of internal or external hemorrhoidal pathology is primarily based on hygiene and dietetic measures and regularization of transit. In the case of external hemorrhoidal pathology, treatment may also include Non-Steroidal Anti-Inflammatory Drugs (NSAIDs) and topical treatment (anesthetic or topical corticosteroid). For internal hemorrhoidal pathology, when these measures are insufficient or when prolapse is present from the outset, instrumental treatment can be offered, allowing the bleeding and / or prolapse to be treated up to grade 3 maximum. This treatment includes sclerosis (less and less practiced), infrared photocoagulation and rubber band ligation. In 10 to 20% of cases, when the prolapse is irreducible, there is anemia of hemorrhoidal origin or the symptoms persist despite well-conducted treatment, surgical treatment may be offered.

The reference surgical technique in France and in Europe is tripedicular hemorrhoidectomy according to the Milligan and Morgan technique, developed at Saint Marks Hospital in London, first published in 1937. It has the advantage of to be the most effective technique, with a low rate of postoperative recurrence and treats both internal and external hemorrhoidal pathology. However, the postoperative period is painful, requires local care and requires cessation of activity for several weeks. On the other hand, there is a risk of potentially serious complications and permanent sequelae: acute retention of urine (2.1-15%), hemorrhage (0.6-5.4%), anal stenosis (6%) , infection (0.5-5%) and anal incontinence (0-6%). Patient selection is essential and contraindicates hemorrhoidectomy in cases of anal incontinence, active suppuration, chronic inflammatory bowel disease, anal intercourse or a history of pelvic radiotherapy.

As an alternative to hemorrhoidectomy, and its painful and restrictive consequences, new minimally invasive surgical techniques that have proven their effectiveness in the treatment of internal hemorrhoidal pathology have emerged over the past twenty years. The two main ones are Longo circular stapling hemorrhoidopexy and Doppler-controlled arterial ligations with mucopexy. Several studies have shown that Longo's hemorrhoidopexy causes less postoperative pain and allows a faster return to activity than after a tripedicular hemorrhoidectomy. On the other hand, the rate of recurrence of hemorrhoidal pathology was higher. This rate was 41% at 12 years and 47.5% at 15 years. In addition, specific and severe complications have been described as rectal perforations, rectovaginal fistulas, perirectal hematomas, pelvic cellulitis, peritonitis and death.

Several comparative studies have shown that arterial ligation under Doppler control with mucopexy was less painful postoperatively than hemorrhoidopexy by circular stapling and that the short- and medium-term efficacy was generally similar. In addition, the postoperative consequences of arterial ligatures under Doppler control with mucopexy seem harmless, with none of the major complications described after stapled hemorrhoidopexy. For these reasons, arterial ligation is now tending to replace hemorrhoidopexy with circular stapling.

The objective of our study is to assess the rate of recurrence of long-term hemorrhoidal pathology in patients who have had arterial ligatures under Doppler control with mucopexy at our center. The results will help guide the practitioner and the patient in the choice of surgical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age is ≥ 18 years
* Patient with hemorrhoidal pathology
* Patient operated, between November 2012 and October 2015, by the technique of arterial ligatures under doppler control with mucopexy
* French-speaking patient

Exclusion Criteria:

* Patient with failure of the technique (defined by the non-reduction in bleeding and / or prolapse scores during the first 3 postoperative months and beyond).
* Patient with a psychiatric pathology likely to influence the follow-up.
* Patient under guardianship or curatorship.
* Patient deprived of liberty.
* Patient under legal protection
* Patient objecting to the use of their data for this research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hemorrhoidal pathology operated, between November 2012 and October 2015, by the technique of arterial ligatures under Doppler control with mucopexy
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2021-02-12 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
Recurrence rate | Months 60
  this outcome corresponds to the cumulative recurrence rate of symptoms of hemorrhoidal pathology, more than 60 months after performing arterial ligations under Doppler control with mucopexy.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent De Parades, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Result] Riss S, Weiser FA, Schwameis K, Riss T, Mittlbock M, Steiner G, Stift A. The prevalence of hemorrhoids in adults. Int J Colorectal Dis. 2012 Feb;27(2):215-20. doi: 10.1007/s00384-011-1316-3. Epub 2011 Sep 20. PMID 21932016
- [Result] van Tol RR, Kleijnen J, Watson AJM, Jongen J, Altomare DF, Qvist N, Higuero T, Muris JWM, Breukink SO. European Society of ColoProctology: guideline for haemorrhoidal disease. Colorectal Dis. 2020 Jun;22(6):650-662. doi: 10.1111/codi.14975. Epub 2020 Feb 17. PMID 32067353
- See also: Recommandations pour la pratique clinique sur le traitement de la maladie hémorroïdaire — https://www.snfcp.org/wp-content/uploads/2017/Recommandations/RPC-maladie-h%C3%A9morro%C3%AFdaire.pdf